CLINICAL TRIAL: NCT04860726
Title: Effects of Myofascial Release and Joint Mobilization Therapy on Pain, Muscle Thickness, Range of Motion and Functional Disability in Non-Specific Low Back Pain
Brief Title: Myofascial Release and Joint Mobilization Therapy in Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rec/Lhr/1104 Waseem
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: Fascia; Range of motion; Ultrasonography; Low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP A (Experimental): Joint mobilization
  Interventions: Other: Joint mobilization
- GROUP B (Experimental): Myofascial release
  Interventions: Other: Myofascial Release
- GROUP C (Experimental): Joint Mobilization & Myofascial release
  Interventions: Other: Joint mobilization & Myofascial Release

INTERVENTIONS:
Other: Joint mobilization — Maitland Mobilization GIII and GIV i. PA Central and unilateral vertebral pressure ii.Transverse vertebral pressure iii. heating pad for 15 minutes
  Arms: GROUP A
Other: Myofascial Release — Myofascial release is a hands-on soft tissue technique that facilitates a stretch into the restricted fascia. A sustained pressure is applied into the restricted tissue barrier; after 90-120 seconds the tissue will undergo histological length changes allowing the first release to be felt. The therapist will follow the release into a new tissue barrier and holds. After a few releases the tissue will become softer and more pliable.
  The middle point of the Lateral raphae of the Thoracolumbarfascia between the posterior musculofascial junction of the Transversus Abdominis will be identified by ultrasonography. Vertical manual pressure will be applied on the middle point of the thoracolumbarfascia for 1 min ii. heating pad for 15 minutes
  Arms: GROUP B
Other: Joint mobilization & Myofascial Release — Maitland Mobilization GIII and GIV i. PA Central and unilateral vertebral pressure ii.Transverse vertebral pressure iii. heating pad for 15 minutes iv. Myofascial release is a hands-on soft tissue technique that facilitates a stretch into the restricted fascia. A sustained pressure is applied into the restricted tissue barrier; after 90-120 seconds the tissue will undergo histological length changes allowing the first release to be felt. The therapist will follow the release into a new tissue barrier and holds. After a few releases the tissue will become softer and more pliable.
  The middle point of the Lateral raphae of the Thoracolumbarfascia between the posterior musculofascial junction of the Transversus Abdominis will be identified by ultrasonography. Vertical manual pressure will be applied on the middle point of the thoracolumbarfascia for 1 min
  Arms: GROUP C

SUMMARY:
Low back pain is a common condition affecting many individuals at some point in their lives. The prevalence of Non-specific low back pain (LBP) is between 4.2% and 19.6%, which is responsible for high treatment costs, sick leave, and individual suffering, in addition to being one of the main reasons for people to seek health care services. LBP prevalence increases linearly from the third decade of life on, until the 60 years of age, being more prevalent in women. This trial will be a prospective, parallel, double blinded, randomized, interventional clinical trial (comparing Myofascial Release and Joint Mobilization therapy). The patients will be screened by researcher and randomly allocated into either experimental groups. After recruitment, the person will be contacted for allocation so that randomization will be secured and concealed. The outcome measure tools for data quantification will be used i.e. Diagnostic Ultrasound Scanner to measure lumbar multifidus and transversus abdominis muscle thickness, pain pressure algometer to measure pain pressure sensitivity and Halo-digital inclinometer to measure range of motion of the lumbar region. A pilot study was done on a sample of 30 with 10 participants in each group. A sample of 84 participants (28 participants in each group) with an attrition rate of 12%, level of significance 5%, margin of error 20% was the output. Patients will be randomly allocated in 3 groups (Group A, Joint mobilization: Group B, Myofascial Release: Group C, both joint mobilization and myofascial release: Common treatment, Heating for 15 minutes). Each group will receive 4 sessions of treatment in 2 weeks' period on Day 1st day 4th, day 8th and day 12th.Data will be collected on Day 1st; Pre and post-treatment, Day 4th, Day 8th,Day 12th; post treatment and after 1 month. Data will be analyzed with SPSS version.26.

Study will be conducted in Al-Razi Healthcare and Riphah Rehabilitation Centre, Lahore, Pakistan. The duration of study will be 18 months after the approval of synopsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 20 to 50 years for non-specific low back pain diagnosed by researcher according to the non-specific low back pain criteria comprising of history and physical examination. Physical examination should be done in different positions as follows

  * Inspect the back for deformities e.g. stooping forward
  * Palpate for muscle guarding, trigger points
  * Lumbar excursion and range of motion
  * Gait
  * Heel and Toe Walking (Inability to walk on heels alone or toes alone signifies significant muscle weakness) • Hip joint range of motion
  * FABER test (Flexion, Abduction and External Rotation)
  * Straight Leg Raising Test (SLR)
  * Cross SLR
  * Neurological examination • Palpate for muscle guarding, trigger points
  * Femoral Extension Test • Straight Leg Raising Test (SLR)
* Both male and female patients will be recruited.
* Patient diagnosis based on clinical assessment and duration of pain.
* People who have not received physical therapy application or exercise regimen for the past 3 months
* Patients suffering with low back pain for less than 3 months. Severity of Pain should be 3 to 7 on NPRS will be included in the study.
* Patients not received analgesics and Non-steroidal anti-inflammatory drugs for previous 1 week.

Exclusion Criteria:

* Patients already diagnosed with any systemic or musculoskeletal pathology e.g. vasculogenic, viscerogenic, neurogenic Low back pain or any history of any recent trauma etc.
* Patients having as severe to extreme findings of low back pain reflecting the patient irritable.
* Any previous surgery or epidural injection treatment or nerve block in the lumbosacral region.
* Females who are pregnant or any recent pregnancy in past 6 months
* Any sensory or motor deficit in the lower extremities.
* Any signs of reg flags; i.e. tumors, constitutional symptoms, integumentary issues, cauda equina syndromes etc. will be excluded.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonography for Muscle thickness | 1 month
  Interpretation will be done according to the images received after ultrasonography. Readings will be done 1st day, 4th,8th,12th,and after one month.
Pain Pressure Algometer | 1 month
  Pai threshold will be measured by applying pain pressure algometer and readings will be measured.Readings will be done 1st day, 4th,8th,12th,and after one month.
Digital Inclinometer for Range of motion | 1 month
  Instrument used for Range of motion.Readings will be done 1st day, 4th,8th,12th,and after one month.
  Normal Ranges: FLEXION : 0-60, EXTENSION: 0-25, LATERAL FLEXION: 0-25, ROTATION :0-18

SECONDARY OUTCOMES:
Numeric pain rating scale | 1 month
  0= no pain 10 = worse pain Readings will be done 1st day, 4th,8th,12th,and after one month.
Sit and Reach test | 1 month
  Excellent: >34-26 cm Good= 34-26 cm Above average: 32-23 Average: 29-20 Below average: 26-17 cm Poor: 23-14 cm V poor: < 21- <12 cm Readings will be done 1st day, 4th,8th,12th,and after one month.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Principal Investigator — Riphah International University; Hafiz Muhammad Waseem Javaid, PhD*, Principal Investigator — Riphah International University; Muhammad Kashif, PhD, Principal Investigator — Riphah International University; Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Al-Razi Healthcare, Lahore, Punjab Province
  - Riphah Rehabilitation Centre, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No